CLINICAL TRIAL: NCT00360386
Title: Assessment of the Best Loading Dose of Clopidogrel to Blunt Platelet Activation, Inflammation and Ongoing Necrosis.
Brief Title: ALBION "Assessment of the Best Loading Dose of Clopidogrel to Blunt Platelet Activation, Inflammation and Ongoing Necrosis"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C_9108
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel

SUMMARY:
* To compare the Kinetics of inhibition of platelet aggregation (aggregometry) and platelet activation (flow cytometry) with different loading doses of clopidogrel
* To evaluate the effect on various parameters of inflammation and necrosis and the safety of these loading doses

ELIGIBILITY:
Inclusion Criteria:

1. Patient hospitalised with ischemic symptoms (onset < 48 hours) and at least one of the following characteristics of NSTEMI:

   * ECG ST or T changes
   * positive troponin
2. Patient treated on admission with 250-500 mg aspirin (oral or IV) and who will receive low dose aspirin (< or = 100 mg daily) from the next day on
3. Patient treated with bid LMWH (indicated dosage for this indication)

Exclusion Criteria:

1. Catheterization scheduled within 24 hours after randomisation
2. Patient presenting an absolute contra-indication to the use of clopidogrel and/or ASA:

   - history of drug allergy to thienopyridine derivatives or ASA
3. Severe uncontrolled hypertension (BP > 180 / 100 despite therapy)
4. Platelet count < 100 000 / mm3
5. Neutrophil count < 1800 / mm3
6. Patient with increased risk of bleeding, such as severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy
7. History of severe systemic bleeding
8. Patient with any contraindication to LMWH
9. Patient treated with clopidogrel within the last 10 days
10. Patient treated with oral anticoagulants or hirudin or planned to receive these products during the hospitalisation period
11. Patient treated with ticlopidine, dipyridamol, NSAIDs (including Cox1 and Cox2 inhibitors), cilostazol, GPIIb IIIa antagonists or planned to receive any of these products within the next 24 hours following randomisation.
12. Patient whose arm venous status is incompatible with an indwelling catheter
13. Patient presenting an evolving cancer
14. Patient with NYHA class IV heart failure
15. Intubated and ventilated patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2004-03; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Maximum intensity of platelet aggregation induced by ADP 5 µmol/L.

SECONDARY OUTCOMES:
Kinetic profile by aggregometry. Kinetic profile of platelet activation by flow cytometry - Inflammation parameters/markers of necrosis. Death, myocardial infarction, ischemic recurrences leading to revascularisation and/or rehospitalisation.Safety.

CONTACTS AND LOCATIONS:
Overall Officials: SAGNARD Luc, Study Director — Sanofi

REFERENCES:
- [Result] Montalescot G, Sideris G, Meuleman C, Bal-dit-Sollier C, Lellouche N, Steg PG, Slama M, Milleron O, Collet JP, Henry P, Beygui F, Drouet L; ALBION Trial Investigators. A randomized comparison of high clopidogrel loading doses in patients with non-ST-segment elevation acute coronary syndromes: the ALBION (Assessment of the Best Loading Dose of Clopidogrel to Blunt Platelet Activation, Inflammation and Ongoing Necrosis) trial. J Am Coll Cardiol. 2006 Sep 5;48(5):931-8. doi: 10.1016/j.jacc.2006.04.090. Epub 2006 Aug 17. PMID 16949482